CLINICAL TRIAL: NCT01651559
Title: A Double Blind Controlled Clinical Trial Comparing The Efficacy Of A Dead Sea Mineral Enriched Body Cream vs Its Carrier as an Adjuvant Treatment For Psoriatic Patients Undergoing Phototherapy
Brief Title: The Efficacy Of A Dead Sea Mineral Enriched Body Cream vs Its Carrier as an Adjuvant Treatment For Psoriatic Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ahava Dead Sea Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: P7BH
Record Dates: First submitted 2012-07-10; First posted 2012-07-27 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Psoriasis Vulgaris
Keywords: modified PASI; narrow band UVB phototherapy; Dead Sea Minerals; Skin auto-Fluorescence; Skin wash samples

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a two-center study aimed to assess the efficacy of Dead Sea Minerals in alleviating symptoms of Psoriasis Vulgaris, in 50 patients undergoing phototherapy. A bilateral left right comparison will be made, after using the study product and the placebo, for 8 weeks, twice daily, on each of the body sides (left right). In addition to the clinical evaluations, skin biochemistry will be studied using non-invasive techniques. The latter will be correlated with the clinical results of the patients. These will serve for future development of diagnostic assays and personalized therapies.

ELIGIBILITY:
Inclusion Criteria:

* Having 2 symetrical (left right)moderate to severe chronic stable plaque type Psoriasis for at least 6 months and candidates for phototherapy treatment

Exclusion Criteria:

* Volunteers with a known allergy to one of the tested materials or to their ingredients.
* Treatment with medication such as anti-inflammatories, anti-histamines, corticosteroids, systemically or topically applied, unless stopped for 4 weeks prior to the trial in the case of systemic treatment and 2 weeks in the case of topical treatment.
* Volunteers in the process of diagnosis or treatment for cancer / kidney disease / liver disease
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers aged 18-70 diagnosed with moderate to severe chronic stable plaque type Psoriasis for at least 6 months and candidates for phototherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
change from baseline of PASI (Psoriasis Area and Severity Index) | 8 weeks
  Grade 2 lesions (left and right- each one assigned a different treatment: study product or placebo)as follows:E=Erythema (redness) I=Induration (thickness) D=Desquamation (scales)
  0 = Absent
  1. = Slight
  2. = Moderate 3= Severe
  4 = Very severe sum the result: modified PASI=E+I+D (in absence of all 3 symptomes the PASI equals 0, if all 3 are very severe then it equals 12.

SECONDARY OUTCOMES:
change from baseline of the Skin Hydration level | 8 weeks
  corneometric measurement of skin capacitance, which indicates hydration level.

CONTACTS AND LOCATIONS:
Overall Officials: Michael David, Professor, Study Chair — Rabin Medical Center
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva